CLINICAL TRIAL: NCT05139602
Title: A Phase 2 Multicenter, Randomized, Double-Blind Placebo-Controlled Study to Evaluate the Safety and Efficacy of Lutikizumab (ABT-981) in Adult Subjects With Moderate to Severe Hidradenitis Suppurativa Who Have Failed Anti-TNF Therapy: Amended Protocol to Include a Lutikizumab Open-Label Sub-study in Subjects Naïve to Biologic Therapy
Brief Title: A Study to Assess Disease Activity and Safety of Subcutaneous Lutikizumab (ABT-981) in Adult Participants With Moderate to Severe Hidradenitis Suppurativa Who Have Failed Anti-Tumor Necrosis Factor (TNF) Therapy and Who Are Naïve to Biologic Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M20-262; 2020-004108-33 (EudraCT Number)
Record Dates: First submitted 2021-11-29; First posted 2021-12-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Lutikizumab; ABT-981
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — lutikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Main Study: Lutikizumab Dose A (Experimental): Lutikizumab Dose A every week
  Interventions: Biological: Lutikizumab
- Main Study: Lutikizumab Dose B (Experimental): Lutikizumab Dose B every other week
  Interventions: Biological: Lutikizumab
- Main Study: Lutikizumab Dose C (Experimental): Lutikizumab Dose C every other week
  Interventions: Biological: Lutikizumab
- Main Study: Placebo (Placebo Comparator): Placebo every week
  Interventions: Drug: Placebo
- Sub-study: Group 1 (Experimental): Period 1: Lutikizumab Dose A every week. Period 2: Lutikizumab Dose A every week.
  Interventions: Biological: Lutikizumab
- Sub-study: Group 2 (Experimental): Period 1: Lutikizumab Dose A every week. Period 2: Lutikizumab Dose A every other week.
  Interventions: Biological: Lutikizumab

INTERVENTIONS:
Biological: Lutikizumab — Subcutaneous Injection
  Other Names: ABT-981
  Arms: Main Study: Lutikizumab Dose A; Main Study: Lutikizumab Dose B; Main Study: Lutikizumab Dose C; Sub-study: Group 1; Sub-study: Group 2
Drug: Placebo — Subcutaneous Injection
  Arms: Main Study: Placebo

SUMMARY:
Hidradenitis suppurativa (HS) is a chronic and often painful inflammatory skin disease which includes the forming of lumps, abscesses and scars in areas of the skin such as under the breasts, under armpits, inner thighs, groin and buttocks. Despite the clinical benefit anti-tumor necrosis factor (TNF) therapy offers to patients with HS, there remains a significant unmet medical need for patients who fail to achieve adequate benefit with anti-TNF therapy. This study will compare lutikizumab (ABT-981) versus placebo for the treatment of adult participants with moderate to severe HS who have failed anti-TNF therapy.

Lutikizumab (ABT-981) is an investigational drug being developed for the treatment of HS. In the Main Study, participants will be put in 1 of 4 groups, called treatment arms. There is a 1 in 4 chance that participants will be assigned to placebo. Around 160 adult participants with moderate to severe HS who have failed anti-TNF therapy will be enrolled in the study at approximately 50 sites worldwide. In the Sub-study, participants will be put in 1 of 2 groups, called treatment arms. Both arms will receive treatment at different dosing intervals. Around 40 adult participants with moderate to severe HS who are naïve to biologic therapy will be enrolled in the study at approximately 20 sites.

In the Main Study, participants will receive subcutaneous injections of lutikizumab (ABT-981) or placebo every week for 16 weeks. In the Sub-study, participants will receive subcutaneous injections of lutikizumab (ABT-981) every week for the first 15 weeks, then either every week or every other week for 36 weeks. There will be an optional Long Term Extension (LTE) for participants who completed Week 52 of the Sub-study and, as confirmed by the investigator, have shown a therapeutic benefit to study drug. Participants would then received lutikizumab using the same assigned dosing regimen as that from Period 2 of the Sub-study for an additional 104 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires and diaries.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of hidradenitis suppurativa (HS) for at least 1 year prior to Baseline as determined by the investigator.
* A total abscess and inflammatory nodule (AN) count of >= 5 at Baseline
* HS lesions must be present in at least 2 distinct anatomic areas.
* Must have failed anti-TNF treatment for HS.
* To be eligible for the Sub-study, participants must be naïve to biologic therapy for treatment of HS.

Exclusion Criteria:

- History of active skin disease other than HS that could interfere with the assessment of HS, including skin infections (e.g., bacterial, fungal, or viral) requiring systemic treatment within 4 weeks of the Baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Hidradenitis Suppurative Clinical Response (HiSCR) | Week 16
  HiSCR is defined as at least a 50% reduction from Baseline in the total abscess and inflammatory nodule (AN) count, with no increase in abscess count and no increase in draining fistula-count relative to Baseline.
Number of Participants with Adverse Events (AEs) | Up to Approximately Week 68
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Numeric Rating Scale (NRS) 30 among Participants with Baseline NRS >=3 | Week 16
  NRS 30 is defined as at least a 30% reduction and at least 1-unit reduction from Baseline in worst skin pain (maximal daily pain), as assessed by the Patient's Global Assessment (PGA) of Skin Pain.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (54):
- United States (25):
  - Medical Dermatology Specialists /ID# 240641, Phoenix, Arizona
  - Mayo Clinic - Scottsdale /ID# 241030, Scottsdale, Arizona
  - Burke Pharmaceutical Research /ID# 240811, Hot Springs, Arkansas
  - UCSF Fresno /ID# 240903, Fresno, California
  - Medderm Associates /ID# 240729, San Diego, California
  - Clinical Trials Research Institute /ID# 240642, Thousand Oaks, California
  - CCD Research, PLLC /ID# 240728, Cromwell, Connecticut
  - Skin Care Research Boca Raton /ID# 240758, Boca Raton, Florida
  - Apex Clinical Trials /ID# 248558, Brandon, Florida
  - GSI Clinical Research, LLC /ID# 240901, Margate, Florida
  - Florida International Rsrch cr /ID# 240902, Miami, Florida
  - Park Avenue Dermatology, PA /ID# 240807, Orange Park, Florida
  - TruDerm Dermatology of Wellington /ID# 240780, Wellington, Florida
  - Dawes Fretzin, LLC /ID# 240701, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center /ID# 240683, Boston, Massachusetts
  - Revival Research Institute, LLC /ID# 241020, Troy, Michigan
  - MediSearch Clinical Trials /ID# 240810, Saint Joseph, Missouri
  - Washington University-School of Medicine /ID# 240797, St Louis, Missouri
  - Advanced Dermatology of the Midlands /ID# 249750, Omaha, Nebraska
  - Duplicate_Skin Specialists, PC /ID# 240804, Omaha, Nebraska
  - Schweiger Dermatology, P.C. /ID# 240900, New York, New York
  - Mount Sinai Doctors Dermatology /ID# 241588, New York, New York
  - Montefiore Medical Center /ID# 240853, The Bronx, New York
  - Essential Medical Research, LLC /ID# 241807, Tulsa, Oklahoma
  - Center for Clinical Studies - Houston (Binz) /ID# 240692, Houston, Texas
- Australia (4):
  - Duplicate_Paratus Clinical Research Woden /ID# 240605, Phillip, Australian Capital Territory
  - Momentum Clinical Research /ID# 240911, Darlinghurst, New South Wales
  - Premier Specialist /ID# 241288, Kogarah, New South Wales
  - Veracity Clinical Research /ID# 241096, Woolloongabba, Queensland
- Canada (5):
  - Beacon Dermatology Inc /ID# 240741, Calgary, Alberta
  - Wiseman Dermatology Research /ID# 240738, Winnipeg, Manitoba
  - Lima's Excellence in Allergy and Dermatology Research Inc /ID# 240814, Hamilton, Ontario
  - Dr. S.K. Siddha Medicine Professional Corporation /ID# 247986, Newmarket, Ontario
  - Dre Angelique Gagne-Henley M.D. inc. /ID# 240739, Saint-Jérôme, Quebec
- Germany (5):
  - Duplicate_Universitaetsklinikum Erlangen /ID# 240872, Erlangen, Bavaria
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 240873, Hamburg, Hamburg
  - Havelklinik /ID# 240874, Berlin, State of Berlin
  - Klinikum Ruhr Univ Bochum /ID# 240870, Bochum
  - Staedtisches Klinikum Dessau /ID# 240871, Dessau
- Greece (5):
  - 401 GSNA - 401 Army General Hospital /ID# 242189, Athens, Attica
  - Duplicate_University General Hospital Attikon /ID# 240371, Athens, Attica
  - General Hospital Andreas Syggros /ID# 241104, Athens, Attica
  - Duplicate_Papageorgiou General Hospital Thessaloniki /ID# 240385, Stavroupoli (Thessalonikis), Thessaloniki
  - General Hospital of Thessaloniki Hippokrateio /ID# 240697, Thessaloniki, Thessaloniki
- Japan (5):
  - Nagoya City University Hospital /ID# 244392, Nagoya, Aichi-ken
  - Fukuoka University Hospital /ID# 244390, Fukuoka, Fukuoka
  - University Hospital Kyoto Prefectural University of Medicine /ID# 244739, Kyoto, Kyoto
  - University of the Ryukyus Hospital /ID# 244848, Nakagami-gun, Okinawa
  - Kindai University Hospital /ID# 245358, Osakasayama-shi, Osaka
- Alma M. Cruz Santana, MD-Private practice /ID# 244514, Carolina, Puerto Rico, Puerto Rico
- Spain (4):
  - Hospital Santa Creu i Sant Pau /ID# 240529, Barcelona, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 240429, Granada, Granada
  - Hospital General Universitario Gregorio Maranon /ID# 240396, Madrid, Madrid
  - Hospital de Manises /ID# 240440, Manises, Valencia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M20-262